CLINICAL TRIAL: NCT03822013
Title: Survey of Miglustat Therapeutic Effects on Neurological and Systemic Symptoms of Infantile Type of Sandhoff and Taysachs Diseases
Brief Title: Effects of Miglustat Therapy on Infantile Type of Sandhoff and Taysachs Diseases (EMTISTD)
Acronym: EMTISTD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The number of controls was insufficient compared to case.
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Mashhad University of Medical Sciences (Other); Kashan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Tavasoli, Principal investigator, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 97-01-30-36953
Record Dates: First submitted 2019-01-22; First posted 2019-01-30 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: GM2 Gangliosidosis; Supportive Care
Keywords: Sandhoff Disease; Tay-Sachs Disease; Miglustat
MeSH Terms: conditions — Gangliosidoses, GM2; Sandhoff Disease; Tay-Sachs Disease | interventions — miglustat

STUDY DESIGN:
Intervention Model Description: Although randomized control trial is the gold standard for clinical trial studies; there are ethical concerns about placebo control group in rare diseases such as Sandhoff and Tay sachs diseases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Miglustat (Experimental): Miglustat is administered, dose is adjusted according to Body Surface Area as below:
  >1.25 : 200 mg TDS 0.88-1.25 : 200mg BID 0.73-0.88 :100mg TDS 0.47-0.73 : 100mg BID <0.47 :100mg daily
  Interventions: Drug: Miglustat
- No Miglustat (No Intervention)

INTERVENTIONS:
Drug: Miglustat — Treatment with Zavesca regimen based on body surface area as follows: SQRT [Height (cm) × Weight (kg)] / 3600 <1.25 : 200mg TDS 0.88- 1.25: 200mg BID 0.73- 0.88: 100 mg TDS 0.47- 0.73: 100 mg BID <0.47: 100 mg Daily
  Other Names: Zavesca
  Arms: Miglustat

SUMMARY:
GM2 gangliosidosis is an autosomal recessive subtype of Lysosomal Storage Diseases in which, Hexosaminidase A-B deficiency is caused by HEXA-B gene. HEXA deficiency is seen in Tay sachs and HEXB deficiency causes Sandhoff disease.

Infantile forms of Sandhoff and Tay sachs are often lethal and management of the patients is supportive including nutrition, hydration, seizure control and management of respiratory problems. Recent studies have suggested new methods of treatment, such as enzyme replacement therapy, bone marrow transplantation and substrate reduction therapy.

The first drug used in SRT was Miglustat. It was introduced in 1980 as an anti HIV agent and later, it was registered under the trademark of Zavesca in 2009 and was used in treatment of Gaucher and Niemann-Pick disease. Zavesca passes blood brain barrier, so causes reduction of cholesterol and glycosphingolipids CNS neurons and relief of neurologic manifestations. Improvements were seen in oculomotor function, cognition, swallowing, motor disturbances and psychological problems after treatment with Zavesca. No effect has been proved on visceral involvement. Weight loss during first year of treatment, diarrhea and dyspepsia are seen as side effects.

Studies on SRT in lysosomal storage disease have different results. Some show improvements in manifestations of Gausche, Sandhoff & Tay sachs disease, while others show no valuable benefit for this method of treatment.

Finding an effective treatment for these chronic diseases can improve quality of life for the patients and their families, and also reduce costs for healthcare services. The controversy persists and more studies are needed for judgment. So this study is done to evaluate the effect of Miglustat therapy in Sandhoff and Tay sachs disease, and is believed to help for further studies in this field.

DETAILED DESCRIPTION:
This study is a case- control, open label clinical trial. Patients are all registered with diagnosis of Sandhoff and Tay sachs, and recruited at children's medical center Tehran-IRAN. Diagnosis is confirmed by enzyme level and genetic tests. Case group receive Miglustat therapy for 1 year and frequently assessed. Patients in control group are also assessed for 1 year without receiving Miglustat.

Patients are evaluated for neurologic examination, seizure, nasogastric tube insertion, aspiration pneumonia and quality of life at the beginning of study and every 3 months. Miglustat is considered as an Orphan drug so clinical trials about this drug are designed small and adjusted to limited population.

Variables in neurologic examination are Muscle tone, Muscular atrophy and contracture. motor function is scored according to "Gross Motor Function Classification System" (GMFCS) and quality of life is assessed by Infant Toddle Quality Of Life (ITQOL) questionnaire, with confirmed validity and stability.

Data gathered during frequent visits is registered in check lists and analyzed with SPSS version 18. Quantitative variables express with mean and standard deviation and qualitative variables with frequency and percentile. Analysis of variance for repeated measurements (ANOVA) and nonparametric freedman are tests using for comparisons of Outcomes. Sample size is calculated by formula for clinical trials with repeated measures.

Miglustat is FDA approved for Gaucher and Niemann pick diseases. All patients fill the informed consent and the nature of the study is explained to them. The information of participants is kept confidential. They are informed about side effects of the drug. If any cases at any time decides to exclude themselves from the study they are free to do so.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and enzymatically suspected infants of Sandhoff (SD)/Tay-Sachs (TSD) diseases followed confirmation by molecular study.

Exclusion Criteria:

* Renal impairment
* Loss of follow up
* Other systemic diseases
* Concomitant drug therapy which may affect neurological system function

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Hospitalization frequency change | Baseline and 4, 8, 12 months after intervention and 1-year without intervention
  Method of measurement is checklist.
Pneumonia aspiration frequency change | Baseline and 4, 8, 12 months after intervention and 1-year without intervention
  Method of measurement is checklist.
Seizure Frequency change | Baseline and 4, 8, 12 months after intervention and 1-year without intervention
  Method of measurement is checklist.
Route of feeding change | Baseline and 4, 8, 12 months after intervention and 1-year without intervention
  Method of measurement is checklist.
motor function change | Baseline and 4, 8, 12 months after intervention and 1-year without intervention
  Method of measurement is checklist.

SECONDARY OUTCOMES:
quality of life change | Baseline and 1year
  A total score is reported according to Pediatric Quality Of Life Inventory Infant Scales. Total score range is between 0-45 and higher values represent worse outcomes.

CONTACTS AND LOCATIONS:
Locations (3):
- Iran (3):
  - Kashan University Of Medical Sciences, Kashan, Isfahan
  - Mashhad University Of Medical Sciences, Mashhad, Khorasan
  - Tehran University Of Medical Sciences, Tehran, Tehran Province

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Jarnes Utz JR, Kim S, King K, Ziegler R, Schema L, Redtree ES, Whitley CB. Infantile gangliosidoses: Mapping a timeline of clinical changes. Mol Genet Metab. 2017 Jun;121(2):170-179. doi: 10.1016/j.ymgme.2017.04.011. Epub 2017 Apr 29. PMID 28476546
- [Background] Villamizar-Schiller IT, Pabon LA, Hufnagel SB, Serrano NC, Karl G, Jefferies JL, Hopkin RJ, Prada CE. Neurological and cardiac responses after treatment with miglustat and a ketogenic diet in a patient with Sandhoff disease. Eur J Med Genet. 2015 Mar;58(3):180-3. doi: 10.1016/j.ejmg.2014.12.009. Epub 2014 Dec 12. PMID 25497207
- [Background] Masciullo M, Santoro M, Modoni A, Ricci E, Guitton J, Tonali P, Silvestri G. Substrate reduction therapy with miglustat in chronic GM2 gangliosidosis type Sandhoff: results of a 3-year follow-up. J Inherit Metab Dis. 2010 Dec;33 Suppl 3:S355-61. doi: 10.1007/s10545-010-9186-3. Epub 2010 Sep 4. PMID 20821051
- [Background] Shapiro BE, Pastores GM, Gianutsos J, Luzy C, Kolodny EH. Miglustat in late-onset Tay-Sachs disease: a 12-month, randomized, controlled clinical study with 24 months of extended treatment. Genet Med. 2009 Jun;11(6):425-33. doi: 10.1097/GIM.0b013e3181a1b5c5. PMID 19346952
- [Background] Wortmann SB, Lefeber DJ, Dekomien G, Willemsen MA, Wevers RA, Morava E. Substrate deprivation therapy in juvenile Sandhoff disease. J Inherit Metab Dis. 2009 Dec;32 Suppl 1:S307-11. doi: 10.1007/s10545-009-1261-2. Epub 2009 Nov 4. PMID 19898952
- [Background] Tallaksen CM, Berg JE. Miglustat therapy in juvenile Sandhoff disease. J Inherit Metab Dis. 2009 Dec;32 Suppl 1:S289-93. doi: 10.1007/s10545-009-1224-7. Epub 2009 Nov 4. PMID 19898953
- [Background] Bembi B, Marchetti F, Guerci VI, Ciana G, Addobbati R, Grasso D, Barone R, Cariati R, Fernandez-Guillen L, Butters T, Pittis MG. Substrate reduction therapy in the infantile form of Tay-Sachs disease. Neurology. 2006 Jan 24;66(2):278-80. doi: 10.1212/01.wnl.0000194225.78917.de. PMID 16434676
- [Background] Jacobs JF, Willemsen MA, Groot-Loonen JJ, Wevers RA, Hoogerbrugge PM. Allogeneic BMT followed by substrate reduction therapy in a child with subacute Tay-Sachs disease. Bone Marrow Transplant. 2005 Nov;36(10):925-6. doi: 10.1038/sj.bmt.1705155. No abstract available. PMID 16151419
- [Background] Jeyakumar M, Norflus F, Tifft CJ, Cortina-Borja M, Butters TD, Proia RL, Perry VH, Dwek RA, Platt FM. Enhanced survival in Sandhoff disease mice receiving a combination of substrate deprivation therapy and bone marrow transplantation. Blood. 2001 Jan 1;97(1):327-9. doi: 10.1182/blood.v97.1.327. PMID 11133779